CLINICAL TRIAL: NCT04774224
Title: A Phase 2, Randomised, Placebo Controlled Study Investigating the Efficacy of Baricitinib in New Onset Type 1 Diabetes Mellitus
Brief Title: Baricitinib in New-onset Type 1 Diabetes
Acronym: BANDIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St Vincent's Institute of Medical Research (Other)
Collaborators: Juvenile Diabetes Research Foundation Australia (Unknown); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SVI-BARI-01
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes
Keywords: newly diagnosed
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: Randomised placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Prior to study initiation, an independent researcher is responsible for generating the randomization schedule. The randomization schedule including treatment group assignment (active or placebo) will be provided to the pharmacists at each one of the study sites. The study pharmacists will conceal the group assignment from study participants, investigators and study staff including the statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Active Comparator): Baricitinib is an oral JAK1/JAK2-selective inhibitor. Dosage: The dose of baricitinib is 1 x 4mg tablet once daily Duration of administration: 48 weeks Mode of administration: Orally, with or without food
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): One placebo tablet once daily for a duration of 48 weeks. Placebo tablets contain lactose monohydrate, microcrystalline cellulose, croscarmellose sodium and magnesium stearate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Participants will take one tablet of study drug per day for 48 weeks, and will be followed up for 48 weeks after study drug treatment has finished. Two-thirds of participants will receive Baricitinib.
  Arms: Baricitinib
Drug: Placebo — Participants will take one tablet of study drug per day for 48 weeks, and will be followed up for 48 weeks after study drug treatment has finished. One-third of participants will receive Placebo.
  Arms: Placebo

SUMMARY:
Type 1 diabetes (T1D) results from the killing of insulin-producing pancreatic beta cells by cells of the immune system. The study aims to slow the progressive, immune-mediated loss of insulin-producing beta cells that occurs after clinical presentation. The investigators have identified a pathway that is important for immune cells to kill beta cells, and a drug that will block this pathway and prevent beta cell death. This drug, baricitinib, is already in clinical use for rheumatoid arthritis, and is currently in clinical trials for other diseases, including childhood autoimmune diseases. It is hypothesized that baricitinib treatment for 48 weeks will preserve beta cell function in children and young adults with recently-diagnosed T1D.

The trial aims to recruit 83 participants aged 10-30 years who have been recently diagnosed with T1D. Two thirds of the participants will be randomly assigned to receive baricitinib, one third will receive placebo. The trial will test if baricitinib can slow the progressive loss of insulin-producing beta cells in these patients. The primary objective is to determine if baricitinib can reduce the loss of meal-stimulated plasma C-peptide, a measure of beta-cell function. Maintaining endogenous insulin in recent-onset T1D improves glucose control and may lead to long-term improvements in glucose and lower rates of serious diabetes complications and death.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 10 and 30 years (inclusive) at screening;
2. Diagnosis of T1D according to ADA criteria within 100 days prior to starting study drug;
3. Islet autoantibody positivity (one or more of: GADA, IA-2A, IAA (assessed within one week of commencing insulin therapy), ZnT8A);
4. Stimulated (peak or 90 min) C-peptide >0.2 nM during a 2-hour MMTT at the screening visit; or random C-peptide result >0.3 nM during the screening period.
5. Participants of childbearing age who are sexually active must agree to use of effective birth control until the end of the study;
6. Be able to read, understand and give written informed consent;
7. Be willing to comply with intensive diabetes management.

Exclusion Criteria:

1. Use of immunosuppressive or immunomodulatory therapies other than inhaled or topical glucocorticoids;
2. Current or past history of deep vein thrombosis or pulmonary embolism;
3. Impaired renal function defined by estimated glomerular filtration rate (according to the CKD-EPI) of < 60 mL/min/1.73 m2;
4. LDL cholesterol >4mmol/l;
5. Elevated liver function tests at screening:

   1. Aspartate aminotransferase 2x ULN
   2. Alanine aminotransferase 2 x ULN;
6. Clinically significant abnormal laboratory parameters at screening including but not limited to:

   1. Hemoglobin < 8 g/L;
   2. White blood cells <2500 cells/µl;
   3. Lymphocyte count <750 cells/µl;
   4. Platelets <50,000 cells/µl;
   5. Neutrophils <1200cells/µL;
7. Known hypersensitivity to baricitinib;
8. Known malignancy with the exception of successfully treated non- metastatic basal cell and squamous cell carcinoma;
9. Pregnancy, a desire for pregnancy, breast feeding, or a desire to father a child during the study;
10. Patients with current or recent (within 12 weeks of screening) clinically significant comorbidity, including clinically serious viral, bacterial, fungal, or parasitic infection. Viral infections include HBV, HCV, EBV, HIV, recent herpes zoster and TB;
11. Treatment with any investigational product within 30 days or 5 half - lives (whichever is longer) prior to baseline visit, or concurrent participation in a clinical trial with an investigational product or device;
12. Experienced any of the following within 12 weeks of screening: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association Stage IV heart failure;
13. Any serious medical condition within the previous 4 weeks which places the participant at an unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study, including, but not limited to, symptomatic cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine, haematological and neurological conditions or psychiatric illness/social situations that would limit compliance with study requirements;
14. Have had any major surgery within 8 weeks prior to screening or will require major surgery during the study that, in the opinion of the investigator would pose an unacceptable risk to the participant;
15. History of chronic alcohol abuse or IV drug abuse or other illicit drug abuse within 2 years prior to screening.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the change from baseline of plasma C-peptide area under the curve (AUC) over 2 hours following a mixed meal. | Measured at 48 weeks post commencement of intervention.

SECONDARY OUTCOMES:
Change from baseline in plasma C-peptide AUC over 2 hours following a mixed meal. | Measured at weeks 12, 24, 72 and 96 post commencement of intervention.
Change from baseline in mean daily insulin use over 7 consecutive days. | Measured during the 2 weeks prior to the assessment at weeks 12, 24, 48, 72 and 96 post commencement of intervention.
Change from baseline in glycosylated haemoglobin (HbA1c) levels. | Measured at weeks 12, 24, 48, 72 and 96 post commencement of intervention.
Number of participants with responder status. Responder status is defined as glycosylated haemoglobin (HbA1c) less than or equal to 6.5 percent and mean daily insulin use less than 0.5 international units per kilogram per day (IU/kg/day). | Measured at weeks 12, 24, 48, 72 and 96 post commencement of intervention.
Change in estimated C-peptide (CPEST) from baseline. CPEST is calculated based on six variable routine measures: disease duration, BMI, insulin dose, HbA1c, fasting plasma C-peptide and fasting plasma glucose. | Measured at weeks 12, 24, 48, 72 and 96 post commencement of intervention.
Continuous glucose monitoring (CGM). | Measured at baseline, 12, 24, 48 and 96 weeks post commencement of intervention.
The composite outcome assessing both the frequency, and when relevant, the severity of all adverse events. | Adverse events will be monitored throughout the entire study duration at weeks 0, 2, 4, 8, 12, 16, 20, 24, 36, 48, 72 and 96.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Kay, Prof, Principal Investigator — SVI
Locations (4):
- Australia (4):
  - Women's and Children's Hospital Adelaide, North Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Children's Hospital Melbourne, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification.
Time Frame: Immediately following publication, and for at least 15 years after the end of the study.
Access Criteria: The data will be made available on a case-by-case basis at the discretion of primary sponsor and only to researchers who have obtained ethical approval to access it.
  Access is subject to approvals by the Principal Investigator, Prof Thomas Kay. Enquiries should be directed to tkay@svi.edu.au.

REFERENCES:
- [Background] Waibel M, Thomas HE, Wentworth JM, Couper JJ, MacIsaac RJ, Cameron FJ, So M, Krishnamurthy B, Doyle MC, Kay TW. Investigating the efficacy of baricitinib in new onset type 1 diabetes mellitus (BANDIT)-study protocol for a phase 2, randomized, placebo controlled trial. Trials. 2022 May 23;23(1):433. doi: 10.1186/s13063-022-06356-z. PMID 35606820
- [Result] Waibel M, Wentworth JM, So M, Couper JJ, Cameron FJ, MacIsaac RJ, Atlas G, Gorelik A, Litwak S, Sanz-Villanueva L, Trivedi P, Ahmed S, Martin FJ, Doyle ME, Harbison JE, Hall C, Krishnamurthy B, Colman PG, Harrison LC, Thomas HE, Kay TWH; BANDIT Study Group. Baricitinib and beta-Cell Function in Patients with New-Onset Type 1 Diabetes. N Engl J Med. 2023 Dec 7;389(23):2140-2150. doi: 10.1056/NEJMoa2306691. PMID 38055252
- See also: Trial website — https://www.svi.edu.au/bandit/